CLINICAL TRIAL: NCT06870149
Title: Does Cognitive Groove (Brought to You by GERAS DANCE) Improve Physical Performance in Community-Dwelling Older Adults With Frailty: A Parallel Randomized Controlled Trial
Brief Title: Cognitive Groove (Brought to You by GERAS DANCE)
Acronym: GERAS DANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Professor, Department of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18231
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Frailty; Frail Older Adults; Frailty in Aging; Frailty Syndrome
Keywords: Frailty; Rehabilitation; Dance
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Groove (GERAS DANCE) (Experimental): Classes will occur twice per week for 3 months. Classes follow a consistent sequence of activities (orientation and socialization [10-mins]; warm-up [5-mins]; structured dance [30-mins]; cool-down [5-mins]; socialization and review of weekly hand-outs for balance exercises [10-mins]. The curriculum schedule includes five foundations and seven routines. Cognitive Groove (GERAS DANCE) foundations emphasize learning the ABCs of movement and increasing participants' confidence to move their bodies forward and backward and side-to-side with improved speed and rhythmicity. Cognitive Groove (GERAS DANCE) routines combine the foundational skills into full choreographed dances to music from the '50s and '60s (e.g., rock and roll, jazz, salsa, cha cha cha, rhythm soul, swing, disco, and Bollywood). Participants will receive an intervention-specific study manual that describes the homework exercises for each week.
  Interventions: Other: Dance Rehabilitation Intervention
- Usual Care (No Intervention): The control arm participants will continue with their usual care and normal activities. They will not receive any intervention during the study but will be given the opportunity to participate in Cognitive Groove (GERAS DANCE) programming after the study.

INTERVENTIONS:
Other: Dance Rehabilitation Intervention — Cognitive Groove (GERAS DANCE) presents a novel approach to increasing or maintaining independence and quality of life by improving physical performance and mobility using reminiscent music and rhythmic movement in a fun, safe environment. Cognitive Groove was designed to meet the complex needs of older adults with frailty. Our pilot quasi-experimental studies have demonstrated Cognitive Groove results in clinically significant improvements in walking speed by 0.1 m/s with enhanced temporal-spatial walking parameters and improved lower extremity function, including balance and chair stands.
  Other Names: Cognitive Groove (GERAS DANCE)
  Arms: Cognitive Groove (GERAS DANCE)

SUMMARY:
The goal of this clinical trial is to determine the effect of a community-based rehabilitation intervention (Cognitive Groove, Brought to you by GERAS DANCE), compared to usual care, on clinical outcomes in community-dwelling older adults living with frailty. The main questions it aims to answer are:

1. In community-dwelling older adults living with frailty, is Cognitive Groove more effective than usual care in improving functional movement, physical performance and strength?
2. In community-dwelling older adults living with frailty is Cognitive Groove more effective than usual care in improving frailty status, fear of falling, balance confidence, mood, cognition, grip strength, activities of daily living, life space mobility, loneliness, and quality of life?
3. As a community-based rehabilitation intervention, is Cognitive Groove a cost-effective intervention embedded within the community for older adults living with frailty after 12-months?

Participants will participate in Cognitive Groove classes twice per week for 3 months or receive no intervention (usual care).

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling aged ≥65 years
* At high risk for mobility disability/functional limitations as assessed by the FRAIL Scale ≥2
* Able to ambulate independently (25 m) with or without an assistive device
* Able to follow two-step instructions
* Medical clearance from referring clinician, or for self-referrals, medical clearance from family physician to safely participate in exercise
* Can arrange transportation to the YMCA up to 2 times per week

Exclusion Criteria:

* Unable to speak or understand English
* Current regular participation in a structured exercise program or receiving active physical therapy services
* Severe cardiac or pulmonary disease
* Unstable angina or heart failure
* Severe osteoarthritis (e.g., awaiting joint replacement)
* Parkinson's disease or other progressive neurological disorder
* Receiving palliative care
* Travel/commitments requiring missing more than two weeks

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Performance | Baseline and 3-months
  Physical function will be assessed with the Short Performance Physical Battery [total score]. Higher scores indicate better physical performance [range 0-12].

SECONDARY OUTCOMES:
Change in Walking Speed | Baseline and 3-months
  Walking speed will be assessed with the 400-m Walk Test [walking speed, m/s]. Faster walking speeds indicate better performance.
Change in Walking Speed | Baseline to 3-months
  Change in walking speed will be assessed by 8-ft walking speed [m/s]. Faster walking speeds indicate better performance.
Change in Functional Mobility | Baseline and 3-months
  Functional mobility will be assessed with the Timed Up and Go (TUG) Test [total time, s]. A higher score indicates a greater falls risk (greater or equal to 12 sec) and lower functional mobility.
Change in Dual Task Ability | Baseline and 3-months
  Dual-task ability will be assessed by the TUG-Cognitive (Dual Task Ability) [total time, s]. Higher time indicates worse performance.
Change in Static Postural Control | Baseline and 3-months
  Static postural control will be assessed by the Single Leg Stance Test [total time, s]. Higher scores indicate better postural control.
Change in Hand Grip Strength | Baseline and 3-months
  Hand grip strength will be assessed with a handgrip dynamometer [kg]. Higher measures indicate higher grip strength.
Change in Cognition | Baseline and 3-months
  Cognition will be assessed with the Montreal Cognitive Assessment [total score]. Higher scores indicate better cognition [range 0-30].
Change in Cognition | Baseline and 3-months
  Change in cognition will be assessed using the Trail Making Test (TMT) [total time, s]. Higher time indicates worse performance.
Change in Cognition | Baseline and 3-months
  Cognition will be assessed using the Digit Symbol Substitution Test (DSST) [total score]. Higher scores indicate better cognition [range 0-100].
Change in Frailty | Baseline and 3-months
  Frailty will be assessed with the Fit-Frailty Index [total score]. Higher scores indicate greater frailty [range 0-1].
Change in Fear of Falling | Baseline and 3-months
  Fear of falling will be assessed by the Falls Efficacy Scale International (FES-I) [total score]. Higher scores indicate greater fear of falling [range 16-64].
Change in Balance Confidence | Baseline and 3-months
  Balance confidence will be assessed by the Activities-specific Balance Confidence (ABC) Scale [total score]. Higher scores indicate higher confidence [range 0-100].
Change in Depression/Mood | Baseline and 3-months
  Depression and mood will be assessed with the Patient Health Questionnaire-9 (PHQ-9) [total score]. Higher scores indicate more depressive symptoms [range 0-27].
Change in Loneliness | Baseline and 3-months
  Loneliness will be assessed by the University of California Los Angeles (UCLA) Loneliness Scale [total score]. Higher scores in indicate higher loneliness [range 20-80].
Change in Basic Activities of Daily Living | Baseline and 3-months
  Activities of daily living will be assessed with the Katz activities of daily living questionnaire [total score]. Lower scores indicate greater impairment [range 0-6].
Change in Instrumental Activities of Daily Living | Baseline and 3-months
  Activities of daily living will be assessed with Lawton instrumental activities of daily living questionnaire [total scores]. Lower scores indicate greater impairment [range 0-8].
Change in Life Space Mobility | Baseline and 3-months
  Life space mobility will be assessed with the Life Space Assessment [total score]. Higher scores indicate a larger life space [range 0-120].
Change in Health-related Quality of Life | Baseline, 3-months, and 12-months
  Health-related quality of life will be assessed using the Health Utilities Index (HUI). Higher scores indicate better health-related quality of life [range 0-1].
Change in Healthcare Utilization | Baseline, 3-months, and 12-months
  Number of emergency room visits and hospitalizations will be recorded. Higher number of visits indicates higher healthcare utilization.
Change in Healthcare Utilization | Baseline, 3-months, and 12-months
  Healthcare services use will be recorded. Higher number of visits, medications, etc., indicates higher healthcare utilization.
Change in Falls | Baseline to 3-months
  Number of falls will be assessed by self-report and electronic health record.
Change in Falls-Related Injuries | Baseline to 3-months
  Number of falls-related injuries will be assessed by self-report and electronic health record.
Change in Mobility | Baseline to 3-months
  Change in mobility will be assessed by the total number of steps taken daily (e.g., Actigraph accelerometer). Higher number of steps indicates greater mobility.
Adherence | Baseline to 3-months
  Class attendance and homework completion will be recorded [total number completed]. Higher class attendance and homework completion indicates greater adherence.

OTHER OUTCOMES:
Individual-level Economic Evaluation | Baseline, 3-months, and 12-months
  Individual-level economic evaluations will be assessed by changes in direct medical costs and effectiveness outcomes (e.g., quality-adjusted life years - QALYs), calculate and compare the incremental cost-effectiveness ratio (ICER) (e.g., $/ QALY gained, $/ a visit averted) against a willingness-to-pay threshold ($50,000/QALY) to show if this program represents good value for money.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, Principal Investigator — McMaster University
Locations (1):
- Geras Centre for Aging Research, St. Peter's Hospital, Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No